CLINICAL TRIAL: NCT01258946
Title: The Relationship Between Epicardial Adipose Tissue Thickness, Insulin Resistance and Plasma Adiponectin Concentrations In Patients With Polycystic Ovary Syndrome
Brief Title: Epicardial Adipose Tissue Thickness in Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Dr. Aydogan Aydogdu, Gulhane School of Medicine
Other Study IDs: 1491-764-10/1539; epicardial adipose tissue (Other: Gulhane SM)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2010-08

CONDITIONS: Epicardial Adipose Tissue Pcos
Keywords: epicardial adipose pcos

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the present study was to search whether epicardial adipose tissue thickness, a predictor of increased cardiovascular risk, increases in PCOS patients or not and, if it does, to analyze the relationship of EATT with insulin resistance, adiponectin and biochemical and anthropometric parameters.

DETAILED DESCRIPTION:
Context: Polycystic ovary syndrome (PCOS) is characterized with chronic oligo/unovulations, hyperandrogenism and insulin resistance. Insulin resistance is mostly attributed to visceral adipose tissue. Epicardial adipose tissue thickness (EATT) is in close relation with atherosclerotic coronary heart disease and its importance in PCOS is not determined yet. Thus, we aimed to clarify EATT in patients with PCOS and compare with healthy matched controls. In addition we searched plasma adiponectin levels to clarify its relationship with EATT in patients with PCOS.

Settings: EATT was determined by echocardiography. Insulin resistance is calculated as HOMA-IR and plasma adiponectin levels were determined with ELISA radioimmunoassay at Gülhane School of Medicine, Ankara, Turkey.

Patients: Patients with PCOS and healthy controls who were similar in body mass index (BMI) and age (p=0.118, p=0.081, respectively) were enrolled in the study after having their written consents.

Results: Mean EATT and HOMA-IR levels were significantly higher (p=0.001, p=0.001, respectively) while plasma adiponectin concentrations were significantly lower (p=0.0032) in patients with PCOS than controls. There was no correlation between plasma adiponectin levels and EATT in subjects (p=0.824). EATT levels were in positive correlation with HOMA-IR, plasma triglyceride concentrations and body mass index (BMI) (p=0.022, p=0.027, p=0.022, respectively). HOMA-IR, triglyceride levels, HDL-Cholesterol, LH/FSH ratio were most powerful determinants of EATT in logistic regression modeling (p=0.016, p=0.021, p=0.049, p=0.039, respectively).

Conclusion: EATT is increased in patients with PCOS in concordance with HOMA-IR level and these findings may reflect the increased risk for atherosclerotic cardiovascular disease in this particular patient group.

ELIGIBILITY:
Inclusion Criteria:

* pcos patients, all of the women had normal thyroid-stimulating hormone and prolactin levels, and subjects without possible ovarian tumors, congenital adrenal hyperplasia

Exclusion Criteria:

* BMI greater than 35 kg/m2, any chronic renal or liver disease

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 45 patients wit pcos and 45 control cases
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Mean EATT and HOMA-IR levels were significantly higher (p=0.001, p=0.001, respectively) while plasma adiponectin concentrations were significantly lower (p=0.0032) in patients with PCOS than controls. | 1 year
  june 2009-june 2010
HOMA-IR, triglyceride levels, HDL-Cholesterol, LH/FSH ratio were most powerful determinants of EATT in logistic regression modeling (p=0.016, p=0.021, p=0.049, p=0.039, respectively) | 1 year
  June 2009-June 2010

SECONDARY OUTCOMES:
Level of plasma adiponectin was lower in patients with pcos. | 1 year
  june 2009- june 2010

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)